CLINICAL TRIAL: NCT01185171
Title: Ph II Trial of Induction Chemotherapy With Carboplatin and Paclitaxel, Followed by Concurrent Chemotherapy/Radiation Therapy With ZD1839 (IRESSA), 5-FU, Hydroxyurea, and Twice-Daily Radiation, Followed by Adjuvant ZD1839 Monotherapy in Patients With Locally Advanced Head & Neck Cancer
Brief Title: Trial of Induction Chemotherapy With Carboplatin and Paclitaxel, Followed by Concurrent Chemotherapy/Radiation Therapy With ZD1839 (IRESSA), 5-FU, Hydroxyurea, and Twice-Daily Radiation, Followed by Adjuvant ZD1839 Monotherapy in Patients With Locally Advanced Head & Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12019A
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer
Keywords: Larynx; Lip; Oral Cavity and Pharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases; Lymphoid Interstitial Pneumonia | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ZD1839 500mg by mouth (po) daily (Experimental): Single arm, two-stage, phase II trial of induction therapy with carboplatin and paclitaxel, followed by ZD1839, 5-FU, hydroxyurea, and hyperfractionated radiotherapy, followed by adjuvant ZD1839 alone.
  Interventions: Drug: ZD 1839 500mg

INTERVENTIONS:
Drug: ZD 1839 500mg — Optional Induction chemotherapy:
  Carboplatin and paclitaxel combination will be administered for 2 cycles of 4 weeks duration each. Paclitaxel: 100 mg/m2 in 500 ml of dextrose 5% in water over 3hrs. Carboplatin: Start after completion of paclitaxel on Day 1 AUC 6 (creatinine clearance [CC] + 25). Administered in 100 ml of normal saline over 30min after completion of paclitaxel.
  Resume chemotherapy C2 on D29. ZD1839: 500mg PO QD from D1 of C1 of chemoradiotherapy, uninterrupted until disease progression. Chemotherapy should be administered during all 5 weeks of radiotherapy. P.M.:Start hydroxyurea at 500 mg PO q 12hrs × 6 days. The first daily dose of hydroxyurea on Days 1 through 5 is given 2 hours prior to the first fraction of daily radiotherapy. P.M.:Start continuous infusion of 5-FU at 600 mg/m2/day × 5D. Days 1 through 5: Radiation therapy is administered twice daily at 150 cGy ZD1839 will be administered from day 1 to 14 of every chemoradiotherapy cycle.

SUMMARY:
The purpose of this study is to explore the activity of ZD1839 added to concurrent chemoradiotherapy and as adjuvant monotherapy in patients with locally advanced head and neck cancer. Activity is described in terms of response rate (complete responses only).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of squamous cell or poorly differentiated carcinomas, or lymphoepithelioma of the nasopharynx.
2. Age 18 years or older.
3. Patients with AJCC (6th edition, 2002) stage III or IV head and neck cancer.
4. Patients with AJCC (6th edition, 2002) stage IV head and neck cancer. presenting with cervical lymph node metastasis of an unknown primary (i.e., TxN2 or TxN3) are also eligible.
5. Prior to entry in the study, the resectability and alternative treatment options for each patient will be determined by a team composed of a head and neck surgeon, a radiation oncologist,and a medical oncologist. Stage determination, optimal local treatment, and its timing according to this protocol will be determined at this evaluation. Each patient will be classified as having resectable or unresectable disease. The unequivocal demonstration of distant metastasis (M1) confers ineligibility.
6. Unidimensionally measurable disease (based on RECIST) is desirable but not strictly required. Individuals who are disease free at baseline after excisional biopsy or node dissection will be considered not evaluable for response assessment but are eligible.
7. No prior or radiotherapy.
8. Prior surgical therapy will consist only of incisional or excisional biopsy and organ-sparing procedures such as debulking of airway-compromising tumors or neck dissection in a patient with an unknown primary tumor.
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%.
10. Patients must have normal organ and marrow function as defined below absolute neutrophil count (ANC) ≥ 1,500/μl platelets ≥ 100,000/μl total bilirubin within normal institutional limits aspartate aminotransferase (AST, SGOT)/ alanine aminotransferase (ALT, SGPT) ≤ 2.5 × institutional upper limit of normal alkaline phosphatase ≤ 2 × upper limit of normal creatinine within normal institutional limits

Exclusion Criteria:

1. Unequivocal demonstration of metastatic disease (i.e. M1 disease).
2. Known severe hypersensitivity to ZD1839 or any of the excipients of this product.
3. Any coexisting malignancy that would increase risk of toxicity, interfere with interpretation of toxicity, or is associated with a median survival of less than 24 months.
4. Concomitant use of phenytoin, carbamazepine, barbiturates, rifampin, phenobarbital, or St.John's Wort.
5. Treatment with an investigational drug within 30 days before Day 1 of trial treatment.
6. Incomplete healing from previous surgery.
7. Pregnancy or breast feeding (women of child-bearing potential). Patients should be advised to use effective contraception as appropriate.
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to paclitaxel, Cremophor EL, carboplatin, 5 FU, or hydroxyurea.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection,symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Patients with clinically significant pulmonary dysfunction, cardiomyopathy, or any history of clinically significant CHF are excluded. The exclusion of patients with active coronary artery disease will be at the discretion of the attending physician.
11. Patients must have no uncontrolled active infection other than that not curable without treatment of their cancer.
12. No patients with severe baseline neurologic deficits (> grade II neuropathy) will be treated with induction chemotherapy.
13. Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-01-27 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, MD, Principal Investigator — The University of Chicago Medical Center
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- See also: The University of Chicago Comprehensive Cancer Center Web page — http://uccrc.uchicago.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2003 to October 2004, 70 patients signed consent at three participating institutions.
Pre-assignment Details: 1 patient withdrew before initiating therapy and was not included in the trial. 10 patients underwent surgery to remove all gross disease before initiating study and were unevaluable for response.
Groups:
- ZD1839 500mg by Mouth (po) Daily: Single arm, two-stage, phase II trial of induction therapy with carboplatin and paclitaxel, followed by ZD1839, 5-FU, hydroxyurea, and hyperfractionated radiotherapy, followed by adjuvant ZD1839 alone.
  Induction chemotherapy: ZD 1839 (250mg/day), two cycles of Paclitaxel (100mg/m2 days 1, 8, 15), Carboplatin (AUC 6, day 1). Concurrent chemotherapy and radiation treatment began 1-2 weeks after induction chemotherapy: 4-5 14 day cycles (5 days of 500 mg of hydroxyurea orally every 12 h, 600mg/m2/d of continuous infusion fluorouracil, and 1.5Gy of radiation twice per day followed by 9 days without therapy.
Period: Induction Chemotherapy
Arm/Group | ZD1839 500mg by Mouth (po) Daily
Started | 59
Completed | 57
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Duodenal Ulcer | 1
Period: Concurrent Chemo and Radiation Treatment
Arm/Group | ZD1839 500mg by Mouth (po) Daily
Started | 69
Completed | 66
Not Completed | 3
Not completed — Death | 3
Period: Maintenance
Arm/Group | ZD1839 500mg by Mouth (po) Daily
Started | 60
Completed | 48
Not Completed | 12
Not completed — Elevated liver transaminases | 3
Not completed — Rush | 2
Not completed — Diarrhea | 1
Not completed — Xerostomia | 1
Not completed — Nausea | 1
Not completed — Comorbid Illness | 2
Not completed — Withdrawal by Subject | 1
Not completed — Disease Recurrence | 1

BASELINE CHARACTERISTICS:
Arm/Group | ZD1839 500mg by Mouth (po) Daily
Number analyzed (Participants) | 69
Age, Continuous [Median (Full Range); unit: years] | 55 [49 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 58
  Race: Black | 10
  Race: Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate Achieved 1 Month After Concurrent Chemotherapy and Radiation Treatment
Description: To explore the activity of ZD1839 added to concurrent chemoradiotherapy and as adjuvant monotherapy in patients with locally advanced head and neck cancer. Activity is described in terms of response rate (complete responses only).
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | ZD1839 500mg by Mouth (po) Daily
Number analyzed (Participants) | 59
Participants | 52
Statistical Analysis 1: Comparison: ZD1839 500mg by Mouth (po) Daily; Test type: Non-Inferiority — The power of the study was conducted as a two-stage, non-inferiority phase II trial with a total sample size of 59 patients to detect a 15% lower rate than 80% achieved with TFHX, with alpha = 0.05 and beta = 0.20. In the first stage, 25 patients were recruited, with a plan to terminate if 16 or less complete responses (CR) were observed. Otherwise, additional 34 patients would be recruited and the treatment would be deemed not inferior to historical if more than 45 CRs were observed; p < 0.01, Binomial test for a proportion — Ho: CR rate = 0.65 vs Ha: CR rate > 0.65; proportion = 0.88, 95% CI 2-sided [0.77 to 0.95]

2. Secondary Outcome: 4 Year Overall Survival
Description: Percentage of patients who survived 4 years or more
Time Frame: 0.3 to 4.7 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | ZD1839 500mg by Mouth (po) Daily
Number analyzed (Participants) | 69
percentage of patients | 74 [62 to 83]

3. Secondary Outcome: 4 Year Progression Free Survival
Description: Percentage of patients who survived without progressive disease 4 years or more
Time Frame: 0.3 to 4.7 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | ZD1839 500mg by Mouth (po) Daily
Number analyzed (Participants) | 69
percentage of patients | 72 [60 to 81]

4. Secondary Outcome: 4 Year Disease Specific Survival
Description: Percentage of patients who did not die by the disease within 4 years
Time Frame: 0.3 to 4.7 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | ZD1839 500mg by Mouth (po) Daily
Number analyzed (Participants) | 69
percentage of patients | 89 [77 to 95]

ADVERSE EVENTS:
Time Frame: The adverse events were collected during the IC and CCRT periods (3 months).
Arm/Group | ZD1839 500mg by Mouth (po) Daily
All-Cause Mortality (participants affected / at risk) | 4/69
Serious Adverse Events (participants affected / at risk) | 17/69
Other Adverse Events (participants affected / at risk) | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZD1839 500mg by Mouth (po) Daily (N=69)
Vomiting (Gastrointestinal disorders) | 1
Mucositis (Gastrointestinal disorders) | 7
Anorexia (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Sudden Death (General disorders) | 1
Death NOS (Cardiac disorders) | 1
Infection (General disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD1839 500mg by Mouth (po) Daily (N=69)
Nausea (Gastrointestinal disorders) | 52 — Nausea
Vomiting (Gastrointestinal disorders) | 37
Mucositis (Gastrointestinal disorders) | 64
Constipation (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 63
Diarrhea (Gastrointestinal disorders) | 29
Fever (General disorders) | 15
Anorexia (Gastrointestinal disorders) | 41
Alopecia (General disorders) | 48
Pain (General disorders) | 61
Neutropenia (Blood and lymphatic system disorders) | 62
Neurotoxicity (Nervous system disorders) | 26
Infection (General disorders) | 8
Dermatitis (Skin and subcutaneous tissue disorders) | 62
Thrombocytopenia (Blood and lymphatic system disorders) | 31
EGFR related rash (Skin and subcutaneous tissue disorders) | 32
Palmar-Plantar Erythrodysesthesia (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT01185171/Prot_SAP_000.pdf